CLINICAL TRIAL: NCT01682525
Title: Ovarian Tissue Cryopreservation for Fertility Preservation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Boston IVF (Other)
Responsible Party: Principal Investigator, David Ryley, MD, Reproductive Endocrinologist, Boston IVF
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N09-454
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: Fertility preservation; Ovarian Tissue; Cryopreservation; Assisted Reproductive Technology
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ovarian tissue cryopreservation (Experimental): The ovarian tissue is cryopreserved and stored at Boston IVF, which is an FDA compliant and American Association of Tissue Banks accredited long term storage facility for reproductive tissue.
  Interventions: Other: Frozen ovarian tissue

INTERVENTIONS:
Other: Frozen ovarian tissue — Use of ovarian tissue cryopreserved and stored at Boston IVF

SUMMARY:
To provide a novel fertility preservation option for patients facing a fertility threatening cancer diagnosis or treatment regimen by establishing an ovarian tissue cryopreservation program. To determine if ovarian tissue cryopreservation provides women with a useful, successful option for fertility preservation

The hypothesis is that ovarian tissue cryopreservation for fertility preservation provides an alternative option for fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy which are likely to result in permanent loss of subsequent ovarian function or diminished fertility
* Have a medical condition or malignancy that requires removal of all or part of one or both ovaries
* Patients may have newly diagnosed or recurrent disease
* Be in good health so as to be able to undergo laparoscopic surgery as determined by history and physical examinations, and consultation with the medical oncologist, reproductive endocrinologist, surgeon and anesthesiologist

Exclusion Criteria:

* Moderate to high-risk of ovarian failure due to treatment
* Documented ovarian metastasis
* HIV or hepatitis (B, C)-positive serology
* Absolute surgical contraindications
* ECOG performance status of 0 or 1
* Pregnancy
* Women with psychological, psychiatric, or other conditions which prevent giving fully informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety | 10 years
  Safety, which will be assessed by tracking the number of minor and major complications of the procedure including the following:
  * Minor: Local infection
  * Major: Blood loss requiring blood transfusion, major infection requiring admission or parental antibiotics, injury to surrounding organs requiring further procedures, hospitalization due to unforeseen operative complication

SECONDARY OUTCOMES:
Efficacy | 10 years
  * Proportion of women who attempt pregnancy
  * Proportion of women who become pregnant and outcome
  * Proportion of women using assisted reproduction after re-implantation or ovarian tissue.
  * Menstrual cyclicity and ovarian reserve in those with and without re-implantation

CONTACTS AND LOCATIONS:
Overall Officials: David Ryley, MD, Principal Investigator — Boston IVF
Locations (2):
- United States (2):
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Boston IVF, Waltham, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.bostonivf.com